CLINICAL TRIAL: NCT00328978
Title: A Canadian, Multicenter, Double-Blind, Randomized, Parallel-Group Study of the Safety, Tolerability, and Efficacy of Treatment With Higher Doses of Quetiapine Fumarate (Seroquel®) Greater Than 800 mg/Day in Schizophrenic or Schizoaffective Subjects.
Brief Title: Seroquel STACK Study in Schizophrenic or Schizoaffective Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DC-990-0165; D1441C00023
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia; Schizoaffective Disorders
Keywords: schizophrenia; schizoaffective disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The purpose of the study is to assess and compare the side effect profile, safety, tolerability and efficacy of schizophrenic or schizoaffective subjects non- or partially- responsive to 800 mg/day of quetiapine treated with either 800 mg/day or more than 800 mg/day of quetiapine during 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Men and women, age 18-65 years with persistent positive or negative symptoms with a PANSS total score of ≥ 70 and < 110 and a Clinical Global Improvement (CGI)- Severity of Illness score of at least 4 (moderately ill) at screening. Subjects may be treated as in- or out-patients. Subjects must give written informed consent.

Exclusion Criteria:

* Subjects with other psychiatric, medical or behavioural comorbid disorder that may interfere with study conduct or interpretation.
* Female of childbearing potential, unless the subject is using a reliable method of contraception
* Subjects with alcohol or psychoactive-substance dependence not in full remission or with significant alcohol or substance abuse in the past 3 months will be excluded.
* Laboratory test results outside the range of reference considered by the investigator to be clinically significant.
* Inability to respect the visit schedule and known intolerance to quetiapine at 800mg/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2003-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of subjects (%) experiencing emergent or a worsening of EPS following treatment of quetiapine 800mg or higher than 800 mg/day in schizophrenic or schizoaffective subjects.

SECONDARY OUTCOMES:
To determine the safety, tolerability and efficacy of treatment with quetiapine in with doses higher than 800 mg/day in schizophrenic or schizoaffective subjects.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Canada Medical Director, MD, Study Director — AstraZeneca
Locations (17):
- Canada (17):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, West Claresholm, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, White Rock, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Sydney, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Verdun, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Honer WG, MacEwan GW, Gendron A, Stip E, Labelle A, Williams R, Eriksson H; STACK Study Group. A randomized, double-blind, placebo-controlled study of the safety and tolerability of high-dose quetiapine in patients with persistent symptoms of schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2012 Jan;73(1):13-20. doi: 10.4088/JCP.10m06194. Epub 2011 Jun 14. PMID 21733490